CLINICAL TRIAL: NCT04316169
Title: Hydroxychloroquine (HCQ) in Combination With Abemaciclib and Endocrine Therapy in HR+/Her 2- Advanced Breast Cancer After a Lead in Dose Escalation Cohort of HCQ and Abemaciclib in Advanced Solid Tumors
Brief Title: Hydroxychloroquine, Abemaciclib and Endocrine Therapy in Hormone Receptor Positive (HR+)/Her 2 Negative Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding and PI leaving institution
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Smitha Menon, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00035701
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Solid Tumor; Advanced Breast Cancer
MeSH Terms: interventions — abemaciclib; Hydroxychloroquine; Fulvestrant; Anastrozole; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Abemaciclib and HCQ 200 mg b.i.d. (Experimental): HCQ will have a dose escalation of a 3 + 3 design.
  Interventions: Drug: Abemaciclib; Drug: Hydroxychloroquine 200 mg
- Abemaciclib and HCQ 400 mg b.i.d. (Experimental): HCQ will have a dose escalation of a 3 + 3 design.
  Interventions: Drug: Abemaciclib; Drug: Hydroxychloroquine 400 mg
- Abemaciclib and HCQ 600 mg b.i.d. (Experimental): HCQ will have a dose escalation of a 3 + 3 design.
  Interventions: Drug: Abemaciclib; Drug: Hydroxychloroquine 600 mg
- Abemaciclib + HCQ (Optimal Dose) + endocrine therapy (Experimental): This group will be divided into two cohorts:
  1. eligible participants who are endocrine therapy naive.
  2. eligible participants who had one prior line of endocrine therapy.
  Interventions: Drug: Abemaciclib; Drug: Hydroxychloroquine 200 mg; Drug: Faslodex; Drug: Anastrazole; Drug: Letrozole; Drug: Hydroxychloroquine 400 mg; Drug: Hydroxychloroquine 600 mg

INTERVENTIONS:
Drug: Abemaciclib — 150 mg b.i.d
  Other Names: Verzenio
Drug: Hydroxychloroquine 200 mg — Dose level: 200 mg b.i.d.
  Other Names: Plaquenil
  Arms: Abemaciclib + HCQ (Optimal Dose) + endocrine therapy; Abemaciclib and HCQ 200 mg b.i.d.
Drug: Faslodex — Cohort B will receive Faslodex.
  Other Names: Fulvestrant
  Arms: Abemaciclib + HCQ (Optimal Dose) + endocrine therapy
Drug: Anastrazole — Cohort A will receive anastrazole or letrozole.
  Other Names: Arimidex
  Arms: Abemaciclib + HCQ (Optimal Dose) + endocrine therapy
Drug: Letrozole — Cohort A will receive anastrazole or letrozole.
  Other Names: Femara
  Arms: Abemaciclib + HCQ (Optimal Dose) + endocrine therapy
Drug: Hydroxychloroquine 400 mg — Dose level: 400 mg. b.i.d.
  Other Names: Plaquenil
  Arms: Abemaciclib + HCQ (Optimal Dose) + endocrine therapy; Abemaciclib and HCQ 400 mg b.i.d.
Drug: Hydroxychloroquine 600 mg — Dose level: 600 mg b.i.d.
  Other Names: Plaquenil
  Arms: Abemaciclib + HCQ (Optimal Dose) + endocrine therapy; Abemaciclib and HCQ 600 mg b.i.d.

SUMMARY:
The hypothesis is that abemaciclib synergizes with autophagy inhibitor hydroxychloroquine (HCQ/ Plaquenil), inducing apoptosis leading to tumor regression.

DETAILED DESCRIPTION:
Part 1: 3+3 dose escalation of HCQ combined with abemaciclib in advanced solid tumors.

Part 2: HCQ at top-dose level from part one is combined with abemaciclib and endocrine therapy in HR+/Her 2- advanced breast cancer (ABC) and divided into two cohorts based on prior exposure to endocrine therapy.

Primary Objective

1. Dose-escalation cohort: To determine safety and tolerability of HCQ combined with abemaciclib.
2. Dose-expansion cohort: To determine safety and tolerability of HCQ combined with abemaciclib and endocrine therapy in HR+/Her2- ABC.

Secondary Objectives

1. To assess the clinical efficacy of HCQ in combination with abemaciclib and hormone blockade in the dose- expansion cohort of advanced ER- positive breast cancer participants.
2. To assess the clinical efficacy of HCQ in combination with abemaciclib in the dose- escalation cohort

ELIGIBILITY:
Eligibility Criteria for Part 1 (Enrollment Criteria for the Dose-Escalation Cohort)

Inclusion Criteria for Dose-escalation Phase

1. Patients with advanced or metastatic cancers who are refractory to standard therapy, relapsed after standard therapy, or who have no standard therapy available that improves progression-free or overall survival by at least three months.
2. Intact G1/S checkpoint in tumor tissue defined by positive-Rb staining and negative-low-molecule weight isoforms of cyclin E (LMWE) with staining done on formalin-fixed paraffin embedded slides from archival tissue or cell blocks.
3. Demonstrate measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)1.1 criterion.
4. Age ≥ 18 years.
5. Estimated life expectancy of three months.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
7. Patients with asymptomatic central nervous system (CNS) metastases not requiring use of corticosteroids will be allowed.
8. Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between the last chemotherapy dose and the first dose of the study drug/s (provided the patient did not receive radiotherapy).
9. Patients who received palliative radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between the end of radiotherapy and the first dose of the study drug/s.
10. Patients must be >/= 3 weeks from major surgery. For biologic/targeted agents, patients must be >/= 5 half-lives or >/= 3 weeks from the last dose (whichever comes first).
11. The patient is able to swallow oral medications.
12. Documented ophthalmic exam within the last 12 months demonstrating no evidence of retinopathy. Patients with retinal changes will be considered for enrollment with written clearance from a board-certified ophthalmologist.
13. The patient must sign informed consent prior to registration.
14. The patient has adequate organ function for all of the following criteria, as defined below.

    Laboratory Value Guidance to Establish Adequate Organ Function

    Hematologic:
    * Absolute Neutrophil Count (ANC) ≥ 1.5 × 109/L
    * Platelets ≥100 × 109/L
    * Hemoglobin ≥8 g/dL (Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.)

    Hepatic:
    * Total bilirubin ≤1.5 × upper limit of normal (ULN)
    * Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.
    * Alanine Aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × ULN

    Renal:

    -Creatinine Clearance ≥30 mL/minute
15. Female subjects must meet one of the following:

    * Postmenopausal for at least one year before enrollment, OR
    * Surgically sterile (i.e., undergone a hysterectomy or bilateral oophorectomy), OR
    * If subject is of childbearing potential (defined as not satisfying either of the above two criteria), agrees to practice two acceptable methods of contraception (combination methods require use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 21 days after the last dose of study agent, OR

      o Agrees to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)
16. Male subjects, even if surgically sterilized (i.e., status postvasectomy), must agree to one of the following:

    * Practice effective barrier contraception during the entire study period and through 60 calendar days after the last dose of study agent, OR o Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria for Dose-escalation Phase

1. Serious concomitant systemic disorder that would compromise the safety of the patient or compromise the patient's ability to complete the study, as determined by the treating physician or the principal investigator (for example, interstitial lung disease, severe dyspnea at rest, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea).
2. Second primary malignancy except most in situ carcinomas (e.g., adequately treated non-melanomatous carcinoma of the skin) or other malignancy treated at least five years previously with no evidence of recurrence.
3. Uncontrolled or symptomatic CNS metastases.
4. Known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency.
5. Taking other commercially available medications, which may theoretically either stimulate or inhibit autophagy; these include calcitriol and chloroquine.
6. Taking medications which may lead to interactions with HCQ, including penicillamine, telbivudine, botulinum toxin, digoxin and propafenone.
7. Must not be taking HCQ at baseline.
8. Females who are pregnant or lactating.
9. Uncontrolled infections including and not limited to active bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, human immunodeficiency virus infection with cluster of differentiation 4 (CD4) counts less than 350 and/or AIDS defining opportunistic illnesses known active hepatitis B [for example, hepatitis B surface antigen positive], patients with hepatitis C antibody with detectable hepatitis C viral load.. Screening tests are NOT required for this criterion.
10. The patient has a marked baseline prolongation of QT/QTc interval >470 millisecond using Fridericia's QT correction formula or a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), sudden cardiac arrest, family history of Long QT syndrome.
11. Patients with symptomatic heart failure, uncontrolled arrhythmia, hypokalemia that does not respond to supplementation
12. Patient receiving treatment with strong and moderate Cytochrome P450, family 3, subfamily A (CYP3A) inducers within seven days prior to the first dose of study drugs.
13. Patient receiving treatment with tamoxifen within seven days prior to the first dose of study drugs.
14. Patient receiving treatment with live vaccines within 30 days prior to the first dose of study drugs.
15. Patients receiving medications including herbal supplements which may prolong the QT interval.

Eligibility criteria- Part 2 (Enrollment criteria for the dose-expansion phase)

Inclusion Criteria

1. Postmenopausal women with HR+/ Her2- advanced breast cancer with endocrine naïve disease will be enrolled in Cohort A. Endocrine naïve patients are defined as advanced breast cancer patients eligible for first-line aromatase inhibitor in combination with cyclin-dependent kinase (CDK) 4 / 6 inhibitor therapy. Prior endocrine therapy in the neoadjuvant or adjuvant setting is permitted if the patient had a disease-free interval of more than 12 months.
2. Postmenopausal women with HR +/ Her 2 -advanced breast cancer with endocrine pretreated disease will be enrolled in Cohort B. Endocrine pretreated patients are defined as advanced breast cancer patients who progressed while receiving endocrine therapy as first-line therapy or who had prior endocrine therapy in the neoadjuvant or adjuvant setting with a disease-free interval of less than 12 months and who are otherwise eligible to receive a combination of Faslodex® and CDK 4 / 6 inhibitor may be enrolled in Cohort B.
3. Intact G1/S checkpoint in tumor tissue defined by positive-Rb staining and negative-low-molecule weight isoforms of cyclin E (LMWE) with staining done on formalin-fixed paraffin embedded slides from archival tissue or cell blocks.
4. Age ≥ 18 years.
5. Men with advanced breast cancer may be enrolled in Cohort A or B if they meet eligibility criteria as above for post menopausal women.
6. Peri or premenopausal women may be enrolled in Cohort A or B, if they are receiving a gonadotropin-releasing agonist and meet eligibility criteria as above for postmenopausal women.
7. Female subjects must meet one of the following:

   * Postmenopausal for at least one year before enrollment, OR
   * Surgically sterile (i.e., undergone a hysterectomy or bilateral oophorectomy), OR
   * If subject is of childbearing potential (defined as not satisfying either of the above two criteria), agrees to practice two acceptable methods of contraception (combination methods requires use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 21 days after the last dose of study agent. Patients receiving Fulvestrant should use effective contraception for one year after last fulvestrant dose OR o Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)
8. Male subjects, even if surgically sterilized (i.e., status postvasectomy), must agree to one of the following:

   1. Practice effective barrier contraception during the entire study period and through 60 calendar days after the last dose of study agent, OR
   2. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)
9. Patients with asymptomatic CNS metastases not requiring use of corticosteroids will be allowed
10. Estimated life expectancy of at least six months.
11. ECOG performance status ≤2.
12. Demonstrates measurable disease as defined by RECIST 1.1 criteria or non-measurable bone-only disease.
13. Documented ophthalmic exam within the last 12 months demonstrating no evidence of retinopathy. Patients with retinal changes will be considered for enrollment with written clearance from a board-certified ophthalmologist.
14. Must sign informed consent prior to registration.
15. The patient has adequate organ function for all of the following criteria, as defined below.

    Laboratory Value Guidance to Establish Adequate Organ Function
    * Hematologic
    * ANC ≥ 1.5 × 109/L
    * Platelets ≥100 × 109/L
    * Hemoglobin ≥8 g/dL (Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.)
    * Hepatic
    * Total bilirubin ≤1.5 × ULN
    * Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.
    * ALT and AST ≤3 × ULN
    * Renal
    * Creatinine Clearance ≥30 mL/minute
16. Patients who previously received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events (CTCAE) grade ≤1) from the acute effects of chemotherapy except for residual alopecia or grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and first dose of the study drug/s (provided the patient did not receive radiotherapy).
17. Patients who received palliative radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of palliative radiotherapy and first dose of the study drug/s.
18. The patient is able to swallow oral medications.

Exclusion Criteria

1. Presence of visceral crisis, lymphangitic spread, leptomeningeal carcinomatosis or inflammatory breast cancer.
2. Prior therapy with a CDK 4/6 inhibitor.
3. Serious concomitant systemic disorder that would compromise the safety of the patient or compromise the patient's ability to complete the study, as determined by the treating physician or the principal investigator (for example, interstitial lung disease, severe dyspnea at rest, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea).
4. Second primary malignancy except most in situ carcinoma (e.g., adequately treated non-melanomatous carcinoma of the skin) or other malignancy treated at least five years previously with no evidence of recurrence.
5. Uncontrolled or symptomatic CNS metastases.
6. Known history of G6PD deficiency.
7. Taking other commercially available medications which may theoretically either stimulate or inhibit autophagy; these include calcitriol and chloroquine.
8. Taking medications which may lead to interactions with HCQ, including penicillamine, telbivudine, botulinum toxin, digoxin, and propafenone.
9. Must not be taking HCQ at baseline.
10. Females who are pregnant or lactating.
11. The patient has active bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]). No screening tests is required for this criterion.
12. The patient has a marked baseline prolongation of QT/QTc interval >470 millisecond using Fridericia's QT correction formula or a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest ,family history of Long QT syndrome.
13. Patients with symptomatic heart failure, uncontrolled arrhythmia, hypokalemia that does not respond to supplementation
14. Patient receiving treatment with strong and moderate CYP3A inducers within seven days prior to the first dose of study drugs.
15. Patient receiving treatment with tamoxifen within seven days prior to the first dose of study drugs.
16. Patient receiving treatment with live vaccines within 30 days prior to the first dose of study drugs.
17. Patients receiving medications, including herbal supplements, which may prolong the QT interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities during dose-escalation phase. | 28 days for each cohort
  The number of participants with dose-limiting toxicities during the dose-escalation phase (HCQ in combination with abemaciclib).
Dose-limiting toxicities in dose-expansion phase. | 28 days for each cohort
  The number of participants with dose-limiting toxicities during the dose-expansion phase (maximum-tolerated dose of HCQ and abemaciclib in combination with endocrine therapy.

SECONDARY OUTCOMES:
Progression-free survival. | 1 Year
  This measure is the number of months participants remain free from evidence of disease. Participants will undergo imaging every eight weeks and results will be reported annually.
Overall response rate. | 1 Year
  The number of participants who have a partial or complete response based on tumor measurement by CT or MRI using RECIST 1.1. Participants will be imaged every eight weeks and reported annually.

CONTACTS AND LOCATIONS:
Overall Officials: Smitha Menon, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No